CLINICAL TRIAL: NCT02117986
Title: Clinical and Microbiological Efficacy and Mortality of a Loading Dose of Colistin in Critical Ill Patients
Brief Title: Efficacy and Mortality of a Loading Dose of Colistin in Critical Ill Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Barros Luco Trudeau (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA13I20317
Record Dates: First submitted 2014-04-02; First posted 2014-04-21 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Gram Negative Bacterial Infections
Keywords: critically ill patients; colistin dosing; multidrug resistant bacteria
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — Colistin; colistinmethanesulfonic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- loading dose of colistin (Experimental): Patients will receive a loading dose of colistin (6 million international units) followed by a maintenance dose of 3 million international units of colistin every 8 hours intravenous
  Interventions: Drug: colistin
- without loading dose of colistin (Active Comparator): Patients will receive 3 million international units of colistin every 8 hours intravenous
  Interventions: Drug: colistin

INTERVENTIONS:
Drug: colistin — One arm will receive a loading dose of colistin (6 million international units), and a maintenance dose of 3 million every 8 hours. The other arm will receive a maintenance dose of 3 million international units every 8 hours.
  Other Names: colistimethate sodium; polymyxin e

SUMMARY:
The study hypothesis is that the loading dose of intravenous colistin (6 million of international units) is associated with greater clinical and microbiological efficacy, and reduced mortality of critically ill patients infected by multidrug resistant Gram- negative bacilli, compared to a scheme without loading dose.

DETAILED DESCRIPTION:
It is a prospective, multicenter, randomized, controlled study to evaluate a scheme with and without a loading dose of 6 million international units of colistin, followed by a maintenance dose of 3 million international units every 8 hours intravenous. The study should be conducted in 3 hospitals in Chile, in critically patients presenting infection by multidrug Gram-negative bacteria and requiring be treated with colistin for at least 48 hours. The objectives of the study are: to evaluate the clinical and microbiological response, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized in critical care units
* patient infected by multi drug resistant Gram negative bacteria susceptibly only to colistin
* source of infection: blood, respiratory, intra abdominal or urinary

Exclusion Criteria:

* pregnant or breastfeeding patients
* patient with a history of hypersensitivity to colistin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with clinical response to treatment | up to 1 week
  remission or reduction of clinical signs of infection
percentage of patients with microbiological response | up to 1 week
  negative culture at the same site where the positive culture was obtained before
mortality | during their stay in the intensive care unit
  the mortality during their stay in the intensive care unit, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Rojas, MD, PhD, Principal Investigator — Hospital Barros Luco Trudeau
Locations (2):
- Chile (2):
  - Hospital Barros Luco Trudeau, Santiago, Santiago Metropolitan
  - Hospital de Puerto Montt, Port Montt